CLINICAL TRIAL: NCT00261300
Title: Long-term Pantoprazole Trial in Patients With Symptoms of Chronic Acid Peptic Complaints
Brief Title: Long-term Pantoprazole Trial in Patients With Symptoms of Chronic Acid Peptic Complaints (BY1023/VMG-708)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/VMG-708
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2008-12

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Peptic Ulcers
Keywords: Gastric acid; GERD; Gastroesophageal reflux disease; Pantoprazole; Proton pump inhibitor
MeSH Terms: conditions — Gastroesophageal Reflux; Peptic Ulcer | interventions — Pantoprazole

ARMS (1):
- 1 (Experimental): Pantoprazole 40 mg
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Long term Pantoprozole trial

SUMMARY:
Gastroesophageal reflux disease (GERD) is a medical condition affecting the stomach and esophagus. GERD might occur when the lower esophageal sphincter does not close properly and stomach contents leaks back (refluxes) into the esophagus. GERD is one of the most common medical disorders, with estimates of up to 50% of adults reporting reflux symptoms. One of the main symptoms of GERD is heartburn. It occurs when the acidic content from the stomach touches the lining of the esophagus, causing a burning sensation in the chest or throat. Proton pump inhibitors such as pantoprazole can relieve symptoms of GERD and peptic ulcers in a large proportion of patients.

Additionally, long-term treatment with proton pump inhibitors may be needed for patients with chronic ulcer disease not caused by H. pylori (H. pylori is a stomach-dwelling bacteria which is often associated with ulcers in the stomach or duodenum).

The aim of the study is to evaluate the long-term effect of pantoprazole in patients with chronic gastric acid-related complaints. The study duration consists of a 5-year treatment period. Pantoprazole will be administered once daily. The study will provide further data on long-term safety, tolerability, and efficacy of pantoprazole.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients who completed ALTANA Pharma study BY1023/FK3006 (long-term clinical trial regarding efficacy and tolerability of Pantoprazole in patients not responding to treatment with H2-receptor antagonists or omeprazole)
* Written informed consent

Main Exclusion Criteria:

* Concomitant diseases
* Pregnant or nursing female patients; female patients of childbearing potential who are not using reliable contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2000-10; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events, laboratory values). | 5 years

SECONDARY OUTCOMES:
Evaluation of gastrointestinal symptoms, histological parameters. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Gorig Brunner, Prof. Dr., Principal Investigator — 30659 Hannover, Germany
Locations (1):
- Altana Pharma/Nycomed, Hanover, Germany